CLINICAL TRIAL: NCT03933644
Title: Comparison of the Ambu Aura GainTM With Gastric Tube Versus the Ambu Aura GainTM Without Gastric Tube in Endontolous Patient
Brief Title: Ambu Aura GainTM Guided vs Non Guided in Edentulous Ambu Aura GainTM Without Gastric Tube in Endontolous Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zahnlos
Record Dates: First submitted 2019-04-04; First posted 2019-05-01 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Oropharyngeal Leak Pressure
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambu Aura Gain TM with gastric tube (Other)
  Interventions: Device: Gastric Tube
- Ambu Aura Gain TM without gastric tube (Other)
  Interventions: Device: No gastric Tube

INTERVENTIONS:
Device: Gastric Tube — SGA is inserted with a gastric tube as guide for insertion
  Arms: Ambu Aura Gain TM with gastric tube
Device: No gastric Tube — SGA is inserted without a gastric tube as guide for insertion
  Arms: Ambu Aura Gain TM without gastric tube

SUMMARY:
The Ambu® Aura GainTM is a relatively new 2nd generation Supraglottic Airway Device (SGA) with a second port, providing gastric access to drain gastric content and air and it has an intergrated bite-block that helps avoiding rotation of the SGA.

It has been described and it is known from daily routine, that SGA in edentulous patient provide inferior oropharyngeal leak pressure (OLP).

The aim of the study is to evaluate if the placement of a gastric tube through the second orifice leads to better OLP and lowers the number of intervention needed for replacing the SGA.

The study also evaluates the OLP after 15 minutes and after 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - 3
* Signed informed consent
* Age 18 - 90 years
* Edentolous (or partial) patients
* Patients scheduled for elective surgery

Exclusion Criteria:

* Patients with a known or predicted difficult airway
* Patients with anatomical disorders in the upper airway, the oesophagus or the trachea
* Patients at risk for aspiration
* Body mass index (BMI) > 40 kg/m2

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal Leak Pressure | immediately after insertion
  after insertion

SECONDARY OUTCOMES:
Oropharyngeal Leak Pressure | 15 minutes
  after 15 minutes
Oropharyngeal Leak Pressure | 30 minutes
  after 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Gasteiger, Dr, Principal Investigator — Departement for Anaesthesia and Intensive Care - Medical University Innsbruck
Locations (1):
- MUInnsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No